CLINICAL TRIAL: NCT03276624
Title: Early Outcome in Chronic Unstable Angina Patients With Low Ejection Fraction After CABG
Brief Title: Early Outcome in Unstable Angina Patients With Low EF After CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Elkhawaga, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABGlowEF
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: CABG in Low EF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with low EF undergoing CABG (Other): Chronic Unstable Angina patients with low ejection fraction and a viable myocardium will undergo surgical revascularization CABG
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — surgical revascularization of stenosed coranary arteries using arterial and venous grafts.

SUMMARY:
Coronary artery bypass grafting (CABG) among patients with reduced myocardial function remains a surgical challenge despite improvement in surgical technique, myocardial protection and postoperative care. Such cases are considered as high risk and associated with a higher peri-operative mortality than those with normal left ventricular function (LVF). Patients with low EF are at higher risks of sudden death, ventricular arrhythmia, and worsening heart failure due to recurrent ischemia. Therefore,early recognition of patients at risk for a worse outcome plays a pivotal role in the decision making process, allowing the prompt institution of an adequate support.

DETAILED DESCRIPTION:
Current treatment options for Chronic Unstable Angina patients with low Ejection Fraction include intensive medical therapy, surgical revascularization, ventricular remodeling, and heart transplantation. Medical treatment alone is problematic because of limited long-term survival. Heart transplantation offers excellent results with a 65.6 % 5-year survival rate; however, the scarcity of donor organs, the need for lifelong immunosuppression and the fact that heart transplantation has been restricted to those without co-morbid medical conditions and relatively restricted to those younger than 65 years of age makes this option impractical for a majority of patients. As a result, coronary artery bypass graft (CABG) surgery is the optimal therapeutic approach and remains superior to medical therapy. Numerous controlled trials of coronary artery bypass grafting in patients with low left ventricular ejection fraction (LVEF), have shown that these are the patients that benefit most from revascularization, especially if symptoms of angina or ischemia are present. This benefit is not only for symptoms, but also on longevity. It is believed that the most important factor for successful surgical recovery may be the viability of revascularized myocardium.

ELIGIBILITY:
Inclusion Criteria:

1. Angiographic indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia.
2. Preoperative EF ≤ 40 %.
3. Preoperative myocardial viability (by cardiac MRI).
4. Willing and able to provide written informed consent and comply with study requirements.
5. Patient is willing to comply with all follow-up visits.

Exclusion Criteria:

1. Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema, cardiogenic shock) at the time of enrollment.
2. Prior surgery with the opening of pericardium.
3. Evidence of non-viable (scarred) myocardium.
4. Prior stroke (within 6 months)or more than 6 months if there are substantial neurological defects.
5. Acute ST-elevation MI within 72 hours prior to enrollment requiring revascularization.
6. Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stenting).
7. Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.
8. Intolerance or contraindication to aspirin or both clopidogrel and ticlopidine.
9. Extra-cardiac illness that is expected to limit survival to less than 5 years e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease.
10. EF ≤ 20 %.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-04 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative Ejection Fraction (EF) | 3 months postoperative
  The EF will be measured 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elminshawy, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospitals, Asyut, Egypt